CLINICAL TRIAL: NCT00194701
Title: Exercise to Improve Sleep in Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sandra Motzer, PhD, University of Washington
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97-4765-D09; HL60042
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Heart Failure
Keywords: heart failure; sleep; exercise; heart rate variability
MeSH Terms: conditions — Heart Failure; Motor Activity

INTERVENTIONS:
Behavioral: Walking exercise

SUMMARY:
Of the more than 2 million Americans with heart failure (HF), up to 70% have disturbed sleep that worsens the dyspnea, fatigue, and reduced daytime function associated with HF. Exercise improves sleep in healthy people but the effects of exercise have not been tested in patients with HF. A controlled, randomized trial is proposed to compare the effects of 16 weeks of usual activity (control) with 16 weeks of regular, supervised walking exercise (treatment), on cardiac function and sleep. Approximately 170 subjects with NYHA Class I, II, or III stable heart failure will be recruited. Subjects in the treatment group will walk for exercise up to 5 times a week for up to 30 minutes.

The purpose of this randomized trial is to examine the effects of 16 weeks of regular walking exercise on cardiac function, sleep, and quality of life in persons with stable New York Heart Association (NYHA) Class I, II or III heart failure.

The specific aims are:

1. To compare the physiologic measures of cardiac function (peak oxygen utilization, exercise capacity, nocturnal arterial oxygen desaturations, and heart rate variability) and self-reported quality of life (i.e., symptoms of dyspnea and fatigue, and the ability to perform activities of daily living) of patients randomized to walking vs. control condition.
2. To compare the somnographic (sleep fragmentation, slow wave sleep, sleep efficiency) and self-reported (sleep effectiveness, sleep disturbance, and nap supplementation) measures of sleep for HF patients randomized to walking vs. control condition.
3. Considering the extent of apnea-hypopnea episodes at study entry and group assignment (walking vs. control), explore whether HF patients with frequent apnea-hypopnea episodes (more than 20 per hour) in the walking group experience greater pretest-posttest improvements in physiologic cardiac and somnographic function, when compared with HF patients with few apnea-hypopnea episodes (less than 20 per hour) assigned to walking, or the control group of HF patients with frequent or few apnea-hypopnea episodes.

HYPOTHESES:

1. Heart failure patients who walk regularly will have better cardiac function than the control group.

   Heart failure patients who walk regularly will have higher self-reported quality of life, less shortness of breath/fatigue, and greater ability to perform activities of daily living than the control group.
2. Heart failure patients who walk regularly will have better sleep than the control group.
3. Heart failure patients with frequent episodes of slowed or stopped breathing during sleep who walk regularly will have a greater improvement in pretest-posttest measures of cardiac function than heart failure patients with few episodes of slowed or stopped breathing during sleep who walk regularly, or the control groups with frequent or few breathing difficulties during sleep.

Heart failure patients with frequent apnea-hypopnea episodes who walk regularly will have a greater improvement (i.e., larger difference) in pretest-posttest somnographic sleep measures of efficient, fragmented, and slow wave sleep, than heart failure patients with few apnea-hypopnea episodes who walk regularly, or the control groups with frequent or few apnea-hypopnea episodes.

DETAILED DESCRIPTION:
PROCEDURES. Walking Exercise Intervention. An individualized program of walking exercise is prescribed (walking up to 5 times a week for up to 30 minutes each session). The protocol for this walking intervention is based on exercise programs adapted from 12 research protocols for patients with NYHA Class II-III heart failure, one cardiac rehabilitation protocol in use for approximately 20 years; and the AHCPR Clinical Practice Guidelines for activity prescriptions for heart failure patients. The walking exercise prescription is based on a modified Naughton treadmill test and a 6-minute walk test, both conducted as part of eligibility screening and used as pretest measures. The target exercise heart rate range is calculated from the peak heart rate (measured on treadmill at the peak of oxygen utilization) minus the resting heart rate, multiplied by 40% to 60%, plus the resting heart rate. Weekly for 6 weeks, and then every other week for 10 weeks, the research nurse makes visits to initiate, monitor, and advance an individualized program of walking exercise.

POPULATION. Our target population was persons diagnosed with heart failure (HF).

Pretest and posttest measures include an exercise tolerance test; two nights of somnographic sleep and oxygen saturation recordings; one 24-hour recording of heart rate variability; and subjective reports of quality of life. One-way analyses of variances (ANOVA) will be used to test for control-treatment group differences in cardiac function (Aim 1) and sleep (Aim 2). Interaction will be examined in a two-way ANOVA of group (HF subjects with frequent vs. few apnea-hypopnea episodes walking vs.control) and time (before and after condition) to determine whether HF subjects with frequent apnea-hypopnea episodes who exercise have better outcomes than HF subjects with few apnea-hypopnea episodes who exercise, or the control group (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Classified by the cardiologist, primary physician, or nurse practitioner as having no dyspnea (shortness of breath, air hunger) at rest but fatigue, dyspnea, or anginal (primarily chest/arm/back/neck) pain or discomfort with either ordinary (New York Heart Association classification, NYHA Class II) or less than ordinary (NYHA Class III) physical activity. They could have been Class I (no symptoms) if they were originally diagnosed as having NYHA Class II or III but had responded to treatment.
* Patients must have had evidence of at least one clinical episode of HF diagnosed by a physician or nurse practitioner as fatigue, shortness of breath, and pulmonary congestion.
* Patients had to have stable HF (defined as no hospitalizations for 3 mos, no medication changes for 1 mo, no dyspnea at rest, and no sustained resting heart rate greater than 95 bpm).

Exclusion Criteria:

Patients were considered ineligible for the study based on the following criteria obtained from the patient's physician or nurse practitioner:

* Diagnosed with Pickwickian syndrome, an extreme variant of sleep apnea characterized by severe obesity, respiratory insufficiency, and bi-ventricular failure;
* Known obstructive sleep apnea;
* Unstable angina, myocardial infarction, or cardiac surgery 3 mos prior to study entry;
* Aortic stenosis;
* Routine use of theophylline;
* Kyphoscoliosis (spinal curvature) to the extent that chest and abdominal bands used in sleep recordings could not be kept in place;
* Receiving antidepressant therapy;
* Cardiac transplant recipient;
* Psychiatric diagnoses of manic depression, dementia, or depression;
* Inability to walk without assistance;
* Inability to speak/read English;
* Known atrial fibrillation;
* Current use of nocturnal continuous positive airway pressure (CPAP) or oxygen therapy; and
* Already participating in an exercise program meeting or exceeding the level of activity in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152
Dates: Start 1998-04; Study Completion 2002-03

PRIMARY OUTCOMES:
Somnographic and self-reported measures of sleep.

SECONDARY OUTCOMES:
Physiologic measures of cardiac function and self-reported holistic and health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Motzer, PhD, RN, Principal Investigator — University of Washington School of Nursing
Locations (1):
- University of Washington, Seattle, Washington, United States